CLINICAL TRIAL: NCT02275611
Title: Oxytocin Treatment of Alcohol Dependence: A Randomized, Placebo-Controlled Trial
Brief Title: Oxytocin Treatment of Alcohol Dependence
Acronym: OT-ETOH2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Cort Pedersen, MD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-1862a
Record Dates: First submitted 2014-02-08; First posted 2014-10-27 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Alcohol Withdrawal; Alcohol Dependence
Keywords: oxytocin; alcohol withdrawal; alcohol dependence; alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal oxytocin spray (Syntocinon Spray) (Active Comparator): TID inpatient; BID outpatient for 12 wks
  Interventions: Drug: intranasal oxytocin spray
- Intranasal Placebo Spray (Placebo Comparator): TID inpatient; BID outpatient for 12 wks
  Interventions: Drug: intranasal oxytocin spray; Drug: Intranasal Placebo Spray

INTERVENTIONS:
Drug: intranasal oxytocin spray — Administration of oxytocin in a nasal spray
  Other Names: Syntocinon Spray
Drug: Intranasal Placebo Spray — Intranasal Placebo Spray
  Other Names: Placebo
  Arms: Intranasal Placebo Spray

SUMMARY:
This study will test in individuals who have alcohol dependence (alcohol addiction) the hypotheses 1) that intranasal oxytocin treatment will decrease withdrawal symptoms during medical detoxification and 2) that intranasal oxytocin treatment for 12 weeks in the outpatient setting will decrease drinking.

DETAILED DESCRIPTION:
Study Design This is a randomized, double blind, placebo-controlled early phase II clinical trial.

Recruitment: The study has 2 phases. The first is testing intranasal treatments (oxytocin [OT], placebo) on alcohol withdrawal (the inpatient phase) and the second is testing intranasal treatments on alcohol drinking, craving and anxiety over 12 weeks in the outpatient setting (the outpatient phase). Subjects for the inpatient phase will only be recruited from patients admitted to Freedom House (FRH, mental health center in Chapel Hill, NC) for medical detoxification from alcohol within the last 36 hours. Subjects for the outpatient phase of the study will be inpatients at FRH or the University of North Carolina (UNC) Hospitals who are near the end of their inpatient stay (medical detoxification has been or is nearly completed). Subjects in the inpatient phase of the study at FRH may continue into the outpatient phase after discharge. Subjects for the outpatient phase will also be heavy drinkers from the community who are screened during an initial outpatient clinic visit.

Patients newly admitted to FRH to treat alcohol withdrawal will undergo a brief screening that includes: 1) a recent and past alcohol use interview (Time Line Follow Back, TLFB) and history of alcohol withdrawal interview; 2) a brief psychiatric interview; 3 ) a score on the 10-item CIWA scale of alcohol withdrawal symptoms; 4) a review of potential medical exclusion criteria including a history of seizures or delirium tremens; 5) a spot urine pregnancy test on all prospective female subjects.

Recruitment into the outpatient phase (treatment of outpatient drinking): Patients who undergo medical detoxification from alcohol will be recruited from FRH or from UNC Hospitals toward the end of their admission for participation in a trial to test the efficacy of intranasal OT vs. placebo treatment on alcohol drinking, alcohol craving and anxiety during a 12-week outpatient treatment period. They will be screened to see if they meet study criteria. These individuals will read and sign the Breath Alcohol Policy that states that if their Breathalyzer reading at the beginning of an outpatient clinic visit is >.08 they will not be assessed at that visit and will not drive themselves home but rather will accept a ride from a family member, friend or a cab driver.

Other individuals will be recruited from the community for participation in the outpatient phase of the study who have responded to a radio ad, a UNC listserve ad, a flyer, have been referred by local clinicians or have otherwise become aware of the study. These prospective subjects will undergo a telephone screening interview. If they appear to meet criteria over the phone, they will be further screened during an outpatient clinic visit. They must sign the Breath Alcohol Policy.

Inpatient Treatment of Withdrawal Protocol and Measures: Subjects who enroll in the study shortly after being admitted to FRH will immediately complete the State portion of the Spielberger State-Trait Anxiety Inventory (SSTAI) and the Penn Alcohol Craving Scale (PACS). This will be followed by self-administration of their first intranasal test dose under supervision of research personnel. These subjects will self-administer additional intranasal test doses at 1 and 3 h after the initial dose and then on the evening of that first day of admission. On subsequent admission days at FRH, subjects will self-administer intranasal test doses 3 times per day. After the first intranasal test dose, blood (15 ml) and urine samples will be obtained from subjects at FRH by research personnel for complete blood count (CBC), electrolytes, blood urea nitrogen (BUN), creatinine, glucose, albumin, liver function tests, urinalysis and urine toxicology which will be transported to and run at the UNC Hospital laboratory.

Between the 1st and 3rd initial intranasal test doses, research personnel will complete a more detailed psychiatric interview. Subjects will also complete the University of Rhode Island Change Assessment Scale to assess their stage of motivation to stop or cut back on their drinking, the Drinker's Inventory of Consequences to assess the spectrum of consequences related to drinking, the Family History of Alcoholism Module to assess family history of alcohol problems, the Patient Health Questionnaire (PHQ) to assess symptoms of depression and a Demographic Questionnaire. During the first 2 inpatient days, vital signs and CIWA scores will be obtained (by FRH personnel) every 4 hours or whenever subjects report or nurses observe the onset of withdrawal symptoms. On the 3rd inpatient day, these measures will be obtained 3 times. And on subsequent inpatient days, these measures will be obtained once each day and whenever withdrawal symptoms increase. Subjects will complete the PACS and the SSTAI prior to administration of the 2nd test dose on each inpatient day starting the day after they enter the study. Blood will be drawn early on inpatient day 3 for electrolyte measurements.

In all subjects participating in the inpatient phase of the study, lorazepam (2 mg), a standard medication to decrease withdrawal symptoms, will be administered by mouth (PO) whenever CIWA scores are ≥ 7. CIWA scores will be repeated 1 h after each lorazepam dose and another dose given if the CIWA score remains ≥ 7. Also, lorazepam (2 mg) will be administered if subjects are found to have any of the following elevated vital signs (even if CIWA scores remain low): pulse > 110; diastolic blood pressure > 100; systolic blood pressure > 160. Vital signs (as well as CIWA) will be repeated 1 h after each lorazepam dose and another dose will be given if any of the elevated measures persist. If a subject's CIWA score remains ≥ 7, pulse remains > 110 or diastolic blood pressure remains > 100 after 8 consecutive lorazepam doses, systolic blood pressure remains > 160 after 3 lorazepam doses, or CIWA scores steadily increase despite receiving 3 consecutive lorazepam doses or dangerous symptoms develop (e.g., the onset of hallucinations), a more aggressive detoxification regimen will be initiated and the subject will be dropped from the study. All patients admitted to FRH for alcohol detoxification receive thiamine, folate and multivitamins supplementation.

Initiating Outpatient Test Treatment: Subjects recruited into the outpatient phase of the study at the end of an inpatient admission for medical detoxification from alcohol will be randomized to a treatment group and begin intranasal test treatment during their first outpatient clinic visit after discharge from FRH or UNC Hospitals. Subjects recruited from the community will be randomized and begin intranasal test treatments at a outpatient clinic visit scheduled shortly after their screening clinic visit if assessments at the latter visit indicate they meet inclusion criteria and not exclusion criteria. Several measures will be obtained at the beginning of the clinic visit when subjects begin self-administration of test treatments: Breathalyzer reading, CIWA rating, TLFB interview assessment of recent alcohol consumption, self-ratings on the SSTAI and PACS. Research personnel will then instruct subjects in intranasal self-administration technique and then observe subjects take their first intranasal test dose. Subjects will be given written instructions on intranasal self-administration technique, cleaning the spray bottle nozzle after each dose, storing spray bottles between doses and contacting study personnel if they have question, difficulty with the self-administration procedure or may be experiencing side effects. At the end of the clinic visit, subjects will take home a 60 ml spray bottle (that ejects 0.1 ml metered dose per insufflation) containing 25 ml of test solution which they will use to self-administer test treatment doses twice daily (6 insufflations/dose).

Outpatient clinic visits during the treatment period: Subjects will have follow-up outpatient clinic visits at weeks 1, 2, 3, 4, 6, 8, 10 and 12 after starting intranasal test treatments. Outpatient visits will take place in the Psychiatry Clinics in the UNC Neurosciences Hospital or the Alcohol and Substance Abuse Program (ASAP) clinic which is located off of the UNC campus on a bus line making it more convenient for participants to commute and park thereby facilitating their compliance with the outpatient portion of the study. To enhance continuity, the first visit will be 2-3 days after the clinic visit during which intranasal test treatments are started. At each clinic visit, a Breathalyzer reading, a CIWA score and vital signs will be obtained, a TLFB interview administered to quantify daily alcohol intake since the last clinic visit, and the SSTAI, PACS and PHQ questionnaires will be completed. Subjects will be given a fresh 60 ml intranasal spray bottle containing 25 ml of test substance at clinic visits every 2 weeks. At each clinic visit, subjects' spray bottles will be weighed to monitor compliance. Their intranasal self-administration technique will be reviewed and, if necessary, subjects will be reinstructed in proper technique. At 4, 8 and 12 weeks, blood will be drawn for CBC, liver functions, electrolytes, BUN, creatinine, and a urine sample will be obtained for drug screening and pregnancy tests on all female subjects.

During each clinic visit, 15 minutes of substance use counseling (Medical Management) will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for the inpatient phase (alcohol withdrawal treatment) of the study

  1. Meeting criteria for DSM-IV (Diagnostic and Statistical Manual-IV-TR) alcohol dependence.

  *2. At least one prior episode of DSM-IV alcohol withdrawal as assessed by SCID Alcohol Dependence Module or scoring > 6 on the CIWA scale since admission to the inpatient unit, or having any of the following elevated vital signs since admission: pulse > 110; diastolic blood pressure > 100; systolic blood pressure > 160.

  3. At least 12 heavy drinking days in the 28 days prior to enrollment in the study. A heavy drinking day is defined as >5 standard drinks for men or >4 standard drinks for women.

  4. Women who are able to conceive children must be on an effective form of birth control such as oral contraceptives, intrauterine devices or the use of condoms with spermicide.

  5. Competency to give valid informed consent as indicated by a) a breathalyzer reading at the time the consent form is signed showing an estimated blood alcohol level (BAL) <.08 gm/dL (the consent process is repeated when the BAL level has dropped to 0.00 gm/dL) and b) ability to understand the written informed consent form demonstrated by correctly answering questions about the contents of the form after reading the consent form without help (this will also determine whether prospective subjects can read and understand the study questionnaires).

  6. Ability to get to appointments either through personal or public transportation.
* Inclusion Criteria for the outpatient phase of the study (treatment of heavy drinking) for prospective subjects screened toward the end of their FRH or UNC inpatient stay The same criteria as those listed above for the inpatient phase of the study apply except for the criteria marked with an asterisk.
* Inclusion Criteria for the outpatient phase of the study for prospective subjects recruited from the community and screened during an initial outpatient clinic visit The same criteria as those listed above for the inpatient alcohol withdrawal treatment phase of the study apply except for having a previous history of alcohol withdrawal (inclusion criterion #2)

Exclusion Criteria:

* Exclusion Criteria for the inpatient alcohol withdrawal treatment phase of the study

  * 1. History of alcohol withdrawal-related seizures, delirium tremens or hallucinations.

    2. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., renal insufficiency, cirrhosis, unstable hypertension, unstable diabetes mellitus, seizure disorder). Clinically significant psychiatric illnesses including any psychotic disorder, bipolar disorder, eating disorder, severe depression, or suicidal ideation.

    3. Other substance dependence disorder with the exceptions of nicotine or caffeine. Substance abuse disorders are not exclusionary.
  * 4. Chronic or subchronic ( >3 days in the week prior to admission or outpatient enrollment) treatment with/consumption of benzodiazepines, barbiturates, anticonvulsants or stimulants.
  * 5. Receipt of >6 mg of lorazepam or any dose of a long half-life benzodiazepine between admission for medical detoxification and beginning participation in the study (i.e., receiving the first intranasal dose of test treatment).

    6. AST or ALT (liver function tests) > 5 times ULN (upper level of normal), bilirubin (liver function test) > 1.5 X ULN, sodium < 132 or > 150 mMol/L, potassium < 3.2 or > 5.3 mMol/L.

    7. Women who are pregnant or breastfeeding. 8. Intent to participate in an additional alcohol treatment program other than Alcoholics Anonymous 9. Court-mandated participation in alcohol treatment or pending incarceration.
* Exclusion Criteria for the outpatient phase of the study (treatment of heavy drinking) for prospective subjects screened toward the end of their FRH or UNC inpatient stay The same criteria as those listed above for the inpatient phase of the study apply except for the criteria marked with an asterisk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersem, M.D., Principal Investigator — University of North Carolina, Chapel Hill

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The numbers of subjects recruited into the withdrawal study alone, outpatient study alone, or both = 13. Some people dropped out of the inpatient withdrawal phase after they completed that phase. Additional participants were added for the second, outpatient phase.
Groups:
- Active Comparator:Intranasal Oxytocin Spray (Syntocinon Spray): Syntocinon Spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks.
  Inpatient Withdrawal
- Placebo Comparator: Intranasal Placebo Spray: Placebo spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks Inpatient Withdrawal
- Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon): 2 daily doses intranasal oxytocin spray for 12 weeks
- Outpatient Treatment Placebo Spray: 2 daily doses intranasal placebo spray for 12 weeks
Period: Inpatient Withdrawal
Arm/Group | Active Comparator:Intranasal Oxytocin Spray (Syntocinon Spray) | Placebo Comparator: Intranasal Placebo Spray | Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon) | Outpatient Treatment Placebo Spray
Started | 5 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Outpatient Drinking
Arm/Group | Active Comparator:Intranasal Oxytocin Spray (Syntocinon Spray) | Placebo Comparator: Intranasal Placebo Spray | Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon) | Outpatient Treatment Placebo Spray
Started | 0 | 0 | 6 | 3
Completed | 0 | 0 | 6 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intranasal Oxytocin Spray (Syntocinon): Syntocinon Spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks intranasal oxytocin spray. Inpatient Withdrawal
- Intranasal Placebo Spray: Placebo spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks intranasal placebo spray. Inpatient Withdrawal
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin Spray (Syntocinon) | Intranasal Placebo Spray | Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon) | Outpatient Treatment Placebo Spray | Total
Number analyzed (Participants) | 5 | 4 | 8 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 8 | 5 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 3 | 2 | 6 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 8 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 2 | 7
  White | 4 | 3 | 5 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 6 | 3 | 9
Clinical Institute Withdrawal Assessment for Alcohol (CIWA) [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Institute Withdrawal Assessment for Alcohol (CIWA) measure is a ten item measure of alcohol withdrawal symptoms. The CIWA total score is the summation of 10 questions, with a range from 0 (little to no withdrawal) to 67 (worse alcohol withdrawal). Population: Only 4 oxytocin recipients and 4 placebo recipients were involved in the study of intranasal treatments on alcohol withdrawal as determined by CIWA scores
  scores on a scale
    number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    (all) | 6.41 (1.45) | 5.57 (1.85) |  |  | 5.99 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Institute Withdrawal Assessment for Alcohol (CIWA) Score
Description: The Clinical Institute Withdrawal Assessment for Alcohol (CIWA) measure is a ten item measure of alcohol withdrawal symptoms. The CIWA total score is the summation of 10 questions, with a range from 0 (little to no withdrawal) to 67 (worse alcohol withdrawal).
Time Frame: Change in scores from before initiation of intranasal test treatment and the first 48 hours after initiation of intranasal test treatments
Population: This assessment was done only in the inpatient withdrawal phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intranasal Oxytocin Spray (Syntocinon Spray): Syntocinon Spray 3-4 doses daily inpatient
  intranasal oxytocin spray: Administration of oxytocin in a nasal spray
- Intranasal Placebo Spray: Placebo spray 3-4 doses daily inpatient
  intranasal oxytocin spray: Administration of oxytocin in a nasal spray
  Intranasal Placebo Spray: Intranasal Placebo Spray
Arm/Group | Intranasal Oxytocin Spray (Syntocinon Spray) | Intranasal Placebo Spray
Number analyzed (Participants) | 4 | 4
units on a scale | -2.76 (1.95) | 1.01 (1.62)

2. Secondary Outcome: Total mg of Lorazepam for Detoxification
Description: Cumulative lorazepam received (2 mg doses)
  After initiation of test treatments, CIWA scores and vital signs were obtained every 4 hours or whenever subjects or staff reported/observed significant increases in symptoms. Lorazepam (2 mg dose) was given if CIWA scores were >7, diastolic blood pressure rose to >120, or heart rate rose to >110. An additional 2 mg was given 1 hour after each lorazepam dose if CIWA scores and/or vital signs remained elevated.
Time Frame: 48 hours after initiation of intranasal test doses
Population: This assessment was done only in the inpatient withdrawal phase.
Measure: Mean (Standard Deviation); unit: cumulative lorazepam doses (mg)
Groups:
- Intranasal Oxytocin Spray (Syntocinon Spray): Syntocinon Spray 3-4 doses daily inpatient
- Intranasal Placebo Spray: Placebo spray 3-4 doses daily inpatient
Arm/Group | Intranasal Oxytocin Spray (Syntocinon Spray) | Intranasal Placebo Spray
Number analyzed (Participants) | 4 | 4
cumulative lorazepam doses (mg) | 2.25 (1.26) | 5.25 (2.5)

3. Secondary Outcome: Change in Percentage Heavy Drinking Days
Description: A heavy drinking day is defined by consumption of 5 or more standard drinks for men, 4 or more standard drinks for women. The outcome measure is the change in percentage of heavy drinking days as determine by the Timeline Followback interview between the baseline 90 day period and the first 4 weeks of intranasal test treatment in the outpatient setting.
Time Frame: 90 days prior to admission and 4 weeks in the outpatient setting
Population: This assessment was done only in the outpatient phase.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days change
Arm/Group | Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon) | Outpatient Treatment Placebo Spray
Number analyzed (Participants) | 6 | 3
percentage of heavy drinking days change | -0.377 (0.28) | -0.972 (0.032)

ADVERSE EVENTS:
Groups:
- Intranasal Oxytocin Spray (Syntocinon Spray): Syntocinon Spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks
  intranasal oxytocin spray: Administration of oxytocin in a nasal spray
- Intranasal Placebo Spray: Placebo spray 3-4 doses daily inpatient; 2 daily doses outpatient for 12 weeks
  intranasal oxytocin spray: Administration of oxytocin in a nasal spray
  Intranasal Placebo Spray: Intranasal Placebo Spray
Arm/Group | Intranasal Oxytocin Spray (Syntocinon Spray) | Intranasal Placebo Spray | Outpatient Treatment Intranasal Oxytocin Spray (Syntocinon) | Outpatient Treatment Placebo Spray
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No